CLINICAL TRIAL: NCT02875275
Title: Liquid or Solid State of Food on Glycaemia, Lipaemia and Insulinaemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore Institute of Food and Biotechnology Innovation (Other Government)
Responsible Party: Principal Investigator, JeyaKumar Henry, Principal Investigator, Singapore Institute of Food and Biotechnology Innovation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2015/01098
Record Dates: First submitted 2016-08-01; First posted 2016-08-23 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-08

CONDITIONS: Diabetes; Cardiovascular Disease
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases | interventions — Glucose; Polymethyl Methacrylate; Coconut Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Glucose Solution only (No Intervention): Control drink containing 50 g carbohydrate
- Glucose with grass jelly solution (Active Comparator): Control drink plus 3.12 g grass jelly powder
  Interventions: Other: Glucose with grass jelly solution
- Glucose with grass jelly (solid) (Active Comparator): Control drink plus 3.12 g grass jelly powder in solid form
  Interventions: Other: Glucose with grass jelly (solid)
- Porridge and juice only (No Intervention): Control breakfast containing 50 g carbohydrate.
- Porridge and juice with coconut oil (Active Comparator): Control breakfast, plus 25g coconut oil
  Interventions: Other: Porridge and juice with coconut oil
- Porridge and juice with coconut oil gel (Active Comparator): Control breakfast, plus 25g coconut oil gel
  Interventions: Other: Porridge and juice with coconut oil gel

INTERVENTIONS:
Other: Glucose with grass jelly solution — 50 g glucose and 3.12 g grass jelly dissolve in water (top up to 200g)
  Arms: Glucose with grass jelly solution
Other: Glucose with grass jelly (solid) — 50 g glucose and 3.12 g grass jelly and 3.12g starch dissolve in hot water (top up to 200g)
  Arms: Glucose with grass jelly (solid)
Other: Porridge and juice with coconut oil — Add instant porridge with hot water with oil. Consume with commercially available orange juice
  Arms: Porridge and juice with coconut oil
Other: Porridge and juice with coconut oil gel — Add instant porridge with hot water with oleogel. Consume with commercially available orange juice
  Arms: Porridge and juice with coconut oil gel

SUMMARY:
This study examines the metabolic effects of 3 possible test meals (Oleogel) and/or 3 possible test meals (Grass Jelly). The participants will have the option to voluntarily choose which study part(s) to participate. This study will be evaluated on 40 healthy Chinese male subjects from the general public over a period of one year.

DETAILED DESCRIPTION:
This study examines the metabolic effects of 3 possible test meals (Oleogel) and/or 3 possible test meals (Grass Jelly). The participants will have the option to voluntarily choose which study part(s) to participate. This study will be evaluated on 40 healthy Chinese male subjects from the general public over a period of one year.

Treatments will be randomized to receive 3 different test meals (Oleogel) and/or 3 different test meals. Randomization means assigning the participants to the test meals by chance, like tossing a coin or rolling a dice.

If the participants take part in this study, the participants will be required to come on 3 non-consecutive days and/or 5 non-consecutive days to evaluate the 3 different test meals (Oleogel) and/or 3 different test meal (Grass jelly) respectively, in random order with a minimum of 1 week between the test sessions. For each session, the participants are required to come between 8:00-9:00am, with each session lasting approximately 3.5 hours to 6.5 hours. The participants would have to come following a 10-12 hour overnight fast. An indwelling catheter will be inserted into a vein in the participants' forearm for the remainder of the test session. The investigators will then take a blood sample from the cannula to measure baseline values. The investigators will also take the participant's capillary blood via finger prick to measure blood glucose concentration. After obtaining the baseline blood samples, the investigator will give the participants the test meal to eat within 10 minutes and fill up a 'liking' questionnaire. Following the meal the investigators will take further blood samples (from the cannula and finger pricks) for the next 10, 20, 30, 45, 60, 90, 120, 150, 180, (treatment 4, 5, 6), 210, 240, 270, 300, 330, 360 minutes (Treatment 1, 2, 3).

The amount of blood that will be collected at every time point will be about 5µL droplet from fingerprick and approximately 5mL of blood from cannulation, the accumulative amount per test session will approximately 50 to 80 ml, and the accumulative amount for the entire study duration will be approximately 240 mL of blood by cannula and finger pricks (Part A) and 150 ml (Part B). The investigators will also ask the participants to answer a questionnaire about measurement of hunger and fullness at the same times the blood samples are taken. The appetite-rating questionnaire consists of 100mm continuous lines anchored at each end with opposing statements for a question asked. The specific questions asked will be: 'How hungry do you feel?', 'How full do you feel?', How strong is your desire to eat?', 'How much food do you think you can eat?' and 'Do you have any preoccupation with thoughts of food right now?'. Using a pen, you would have to make a mark on the line corresponding to how you feel.

In addition to the VAS scales, the current trial will collect information on the prospective portion that participants would like to consume for a range of different foods at different time points; at every 30 minutes interval from baseline till the end of each test session. This computer based task presents a range of foods to participants and asks "how much of this food would you like to consume right now?", allowing the participants to move between a series of different portions of each food and select the one that the participants would like to consume at that time based on the participants' feeling of hunger, fullness and desire to eat. The foods will be deliberately chosen to represent common Singaporean meals, desserts and snack foods that are regularly eaten to relieve hunger in different situations and the range of portions available is the same across all foods (20-1200 kcals in 20 kcal steps).

On the evenings before the test sessions, the participants will be expected to come and collect a standard dinner meal. The participants will be advised not to take part in any strenuous physical activities for at least 3 days and avoid caffeine and alcohol consumption the day before the test sessions.

Subjects participation in the study will last a maximum of 20.5 hours (Part A) and 11.5 hours (Part B), include one screening visit lasting around 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* 21-40 years
* Body Mass Index 18-25 kg/m2
* Body weight more than or equals to 45kg
* Normal blood pressure (≤140/90) and normal fasting blood glucose (<6.0 mM)

Exclusion Criteria:

* Have major chronic disease such as heart disease, cancer or diabetes mellitus, intolerances or allergies to test products
* User of insulin or drugs known to affect glucose metabolism and body fat distribution
* People with a major medical or surgical event requiring hospitalization within the preceding 3 months
* Individuals with the presence of disease or drugs which influence digestion and absorption of nutrients
* Current smokers
* People who are on any therapeutic diet/drug

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-27 (Actual)

PRIMARY OUTCOMES:
Change in postprandial blood glucose over 180 minutes period | 180 minutes
  Blood obtained through fingerprick, analysed using Hemocue analyser. Capillary blood glucose will be assessed at 0, 15, 30, 45, 60, 90, 120, 150, 180 minutes.
Change in postprandial plasma triglyceride over 360 minutes period | 360 minutes
  Venous blood obtain through cannula, analysed using Cobas analyser. Venous plasma triglyceride will be assessed at 0, 10, 20, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360 minutes.

SECONDARY OUTCOMES:
Change in postprandial plasma insulin over 360 minutes period | 360 minutes
  Venous blood obtain through cannula, analysed using Cobas analyser. Venous plasma insulin will be assessed at 0, 10, 20, 45, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: JeyaKumar Christiani, Phd, Principal Investigator — Clinical Nutrition Research Centre
Locations (1):
- Clinical Nutrition Reseach Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No